CLINICAL TRIAL: NCT06823648
Title: 23002, Clinical Precision and In-use Analyte Stability Study for 19 Parameters in Adult Arterial Whole Blood for PICO70 and SafePICO
Brief Title: Clinical Precision and In-use Analyte Stability Study for 19 Parameters in Adult Arterial Whole Blood for PICO70 and SafePICO
Status: Completed | Type: Observational
Sponsor: Radiometer Medical ApS (Industry)
Responsible Party: Sponsor
Other Study IDs: DC-086204
Record Dates: First submitted 2024-11-19; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-11

CONDITIONS: Precision and Stability in Adult Arterial Whole Blood Contained in PICO70 and SafePICO for Each Parameter

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Arterial blood samples collected and destroyed immediately after measurements.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adult patients, critically ill and 18 years or older: One single group is included in the study for the investigation of the PICO70 and safePICO syringes.
  Interventions: Device: Arterial blood samplers with needles PICO70 and safePICO syringes

INTERVENTIONS:
Device: Arterial blood samplers with needles PICO70 and safePICO syringes — PICO70 is a self-filling syringe for sample volumes in the range of 0.3-1.5 mL. All syringes are delivered with needle cube for safe needle disposal and a standard tip cap to reduce the risk of blood contact during blood mixing and sample transportation. safePICO is a more advanced group of syringes based on the PICO70 family. They contain a gold coated magnetic steel ball facilitating automatic mixing of the blood when being used with the Radiometer ABL 90 with mixing module. The safePICO is a self-filling syringe covering a volume range of 0.7-1.5 mL and includes a vented safe tip cap (VTC), which simplifies removal of air bubbles and avoid the operator to get in contact with the blood, after attachment to the syringe. Some variants of safePICO are delivered with a needle shield device (NSD) to ensure safe removal of the needle.

SUMMARY:
The purpose is to characterize the precision and in use stability of 19 parameters (pH, pCO2, pO2, cNa+, cCa2+, cCl-, cK+, cGlu, cLac, cUrea/BUN, cCrea, ctHb, sO2, FMetHb, FCOHb, FO2Hb, FHHb, FHbF & ctBil) in arterial blood drawn and stored in self-filling syringes (PICO70 and safePICO) across different lots of samplers measured on ABL90 FLEX PLUS analyzer.

The study aims to determine the total (within Lot and Lot-to-Lot) precision for the PICO70/safePICO in arterial whole blood. Furthermore, the study aims to determine the stability for up to 45 min. at room temperature (18-25 °C) for arterial blood sample analysis in the PICO70/safePICO for all 19 parameters.

DETAILED DESCRIPTION:
The study is a Post-Market Clinical Follow-up (PMCF) randomized unblinded study, expected to be conducted at two sites in Denmark using arterial whole blood samples collected from adult patients to determine the precision and stability for the PICO70/safePICO syringes when measuring 19 parameters (pH, pCO2, pO2, cNa+, cCa2+, cCl-, cK+, cGlu, cLac, cUrea/BUN, cCrea, ctHb, sO2, FMetHb, FCOHb, FO2Hb, FHHb, FHbF & ctBil) using the RMED ABL90 FLEX PLUS analyzer. The 19 parameters will be analysed for each syringe in the syringe series on the ABL90 FLEX PLUS analyzer. For PICO70: Approximately 40+4 (4 contrived sample series) completed series of arterial blood samples consisting of 6 syringes: The syringes will be from three different lots (A,B,C) and analyzed at four different time points, T0, T15, T30 and T45. For safePICO: Approximately 40+4 (4 contrived sample series) completed series of arterial blood samples consisting of 6 syringes: The syringes will be from three different lots (A,B,C) and analyzed at four different time points, T0, T15, T30 and T45. According to guidelines (CLSI GP34) samples should be distributed throughout the analytical measurement range of measurands evaluated. To ensure coverage of the full range for each parameter, it may be necessary to contrive some sample series.

ELIGIBILITY:
Inclusion Criteria:

Subject must be 18 years of age or older. Subject must have an arterial catheter line established as part of the standard of care.

Subject must be suitable for the study according to the protocol evaluated by the principal investigator or designee.

Exclusion Criteria:

Subject is unconscious or otherwise incapable of understanding and signing the informed consent form.

Subject must not have been previously enrolled into this study. Subject must not be known with pregnancy or breastfeeding.

Subject must not be taking the following medications within 72 hours prior to the sample collection:

Acetylsalicylic Acid Sodium Salt at dose equal or above 1 gram/day. Acetylcysteine drug used against paracetamol intoxication. Fluorescein dye (used for the diagnosis of ocular disease). Patent Blue dye (used to mark the lymphatic vessels, arterial territories, and lymph nodes prior to a biopsy).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients 18 years or older, critically ill, but still able to understand and sign the informed consent form and admitted to the hospital having an arterial catheter line established as part of standard of care to minimize the risk to the patient when having blood samples drawn.
  To reach reportable concentrations of the 19 parameters covering the reportable range as much as possible the subject will be a patient in the intensive care unit or another unit corresponding to the emergency care.
Sampling Method: Probability Sample
Enrollment: 63 (Actual)
Dates: Start 2024-06-18 (Actual); Primary Completion 2024-10-28 (Actual); Study Completion 2024-10-28 (Actual)

PRIMARY OUTCOMES:
Precision in adult arterial whole blood in PICO70 and safePICO syringes for each parameter. | One subject delivers blood samples to be measured over time (45 min.)
  The objective is to determine the total (within-lot and between lots) precision for four (19) parameters (pH, pCO2, pO2, cNa+, cCa2+, cCl-, cK+, cGlu, cLac, cUrea/BUN, cCrea, ctHb, sO2, FMetHb, FCOHb, FO2Hb, FHHb, FHbF & ctBil) in arterial blood.
In-use analyte stability in adult arterial whole blood in PICO70 and safePICO syringes for each parameter, measuring at four testing timepoints, T0, T15, T30 and T45. | One subject delivers blood samples to be measured over time (45 min.)

CONTACTS AND LOCATIONS:
Overall Officials: Theis Skovsgaard Itenov, MD, PhD, Principal Investigator — Bispebjerg Hospital, Itensiv afsnit
Locations (1):
- Bispebjerg Hospital, Itensiv afsnit, København NV, Denmark

IPD SHARING:
Plan to Share IPD: Yes
The study results will be available to participating Investigators. The results are also available for supporting the safety and performance of the arterial blood syringes with needles, PICO70, safePICO70 and safePICO self-fill according to requirements.
Supporting Information: CSR
Time Frame: 4 months in Q4 2025 - Q1 2026.